CLINICAL TRIAL: NCT07227545
Title: High Intensity Alternating Current Stimulation as a Neuromodulation Therapy for Alcohol Use Disorder: A Pilot Study
Acronym: HITACS-AUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDu-016
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: High-Intensity Transcranial Alternating Current Stimulation, Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HI-tACS (Experimental): A 40-minute 15mA transcranial alternating current stimulus intervention with 77.5 Hz of real stimulus is conducted twice a day (at least 3 hours apart) for a total of 10 days in the intervention group of AUD.
  Interventions: Device: HI-tACS

INTERVENTIONS:
Device: HI-tACS — A 40-minute 15mA transcranial alternating current stimulus intervention with 77.5 Hz of real stimulus is conducted twice a day (at least 3 hours apart) for a total of 10 days in the intervention group of AUD.

SUMMARY:
This study aims to explore the efficacy of high intensity transcranial alternating current stimulation on individuals with alcohol use disorders. Utilizing a one-arm pilot study design, participants will undergo transcranial alternating current stimulation.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is become a major social and public health problem in China. Craving for alcohol and compulsive drinking behavior are the main symptom of AUD. Previous studies have demonstrated the relationship between cognitive dysfunction and prefrontal-ventral striatum pathway. Studies have shown that abnormal phase synchronization and phase-amplitude coupling (PAC) induced the impairment of cognition, and High-Intensity transcranial Alternating Current Stimulation (HI-tACS) could improve executive-control function thus by adjusting the abnormal synchronization. However, it has not been verified among AUD patients. The investigators assume that tACS could improve AUD patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. This study intends to test the effect of HI-tACS treatment. Three-month follow-up assessment will be conducted to test the changing of the craving and alcohol use behavior. This study will provide a practical and theoretical basis for developing a novel treatment for AUD.

ELIGIBILITY:
Inclusion Criteria:

* Education level of junior high school or above, capable of completing questionnaires and behavioral tests;
* Aged 18-60 years;
* Meet DSM-5 diagnostic criteria for Alcohol Use Disorder;
* No abnormal findings on physical examination;
* Agree to participate in follow-up assessments;
* No contraindications for MRI scanning.

Exclusion criteria:

* Have impaired intelligence (Intelligence Quotient<70);
* Prior tDCS or TMS treatment within the past 3 months;
* Contraindications for TMS therapy (e.g., intracranial metal implants, history of traumatic brain injury, skull defects, cardiac pacemakers, cardiovascular diseases, or epilepsy);
* Severe somatic diseases or major organ dysfunction;
* Psychiatric disorders per DSM-5 criteria (e.g., schizophrenia, schizoaffective disorder, intellectual disability, autism spectrum disorder, dementia, memory impairment, or other cognitive disorders).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of alcohol craving | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Alcohol craving will be measured by the alcohol craving Visual Analog Scale (VAS). The total score of VAS ranged from 0 to 10, in which higher scores mean a higher level of alcohol craving.
The change of drinking behavior | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Questions including monetary loss, time, frequency and interval of drinking will be answered by patients to quantify their gambling behavior.

SECONDARY OUTCOMES:
The change of drinking urge | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Alcohol craving will be assessed using the Alcohol Urge Questionnaire (AUQ). The total score of AUQ ranges from 8 to 56, with higher scores indicating stronger urges to consume alcohol.
The change of abstinence symptom | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Alcohol withdrawal symptoms will be evaluated using the Clinical Institute Withdrawal Assessment for Alcohol, revised version (CIWA-Ar). The total score of CIWA-Ar ranges from 0 to 67, where higher scores indicate more severe alcohol withdrawal symptoms.
Change of the compulsive drinking behavior | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Compulsive drinking behavior will be measured by the short form of the Obsessive-Compulsive Drinking Scale (OCDS). The total score of OCDS ranges from 0 to 40, with higher scores reflecting greater obsessive-compulsive thoughts and behaviors related to alcohol use.
Side effects of the modulation | Immediately after the intervention
  Side effects will be assessed using the Treatment Emergent Symptom Scale (TESS). The scale evaluates the presence and severity of adverse reactions, with higher scores indicating more significant side effects.
Change of depressive symptoms. | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Depressive symptoms will be measured using the 17-item Hamilton Depression Rating Scale (HAMD-17). The total score ranges from 0 to 52, with higher scores indicating more severe depressive symptoms.
Change of anxiety symptoms | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Anxiety symptoms will be assessed using the 14-item Hamilton Anxiety Rating Scale (HAMA-14). The total score ranges from 0 to 56, where higher scores reflect greater anxiety severity.
Change of the sleep quality | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Change of the self-control ability | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Self-control ability will be measured using the Self-Control Scale (SCS). Higher scores of SCS indicate better self-regulation and impulse control.
Change of the risky decision-making performance | Baseline, two weeks after the intervention.
  Risky decision-making performance will be assessed using the Balloon Analogue Risk Task (BART). Higher average pumps in the BART indicate greater risk-taking propensity. Feedback-related negativity (FRN) will be recorded using electroencephalography (EEG), with larger amplitude typically reflecting enhanced sensitivity to negative feedback.
  Pig dice game will be administered during functional magnetic resonance imaging (fMRI) scanning to assess risk-taking decision-making. Higher frequency of continued dice rolls indicates greater risk propensity. Neural activity in the prefrontal cortex and striatum will be analyzed, with increased activation typically associated with risk evaluation and reward processing.
Change of the inhibitory control performance | Baseline, two weeks after the intervention.
  Stop-signal task (SST) will be employed to measure inhibitory control. Longer stop-signal reaction times (SSRT) indicate poorer response inhibition. The N2/P3 components will be recorded using electroencephalography (EEG), with enhanced N2 amplitude and reduced P3 amplitude typically reflecting greater cognitive conflict and inhibitory processing efficiency, respectively.
Change of the resting state neural activity. | Baseline, two weeks after the intervention.
  Resting-state functional magnetic resonance imaging (rsfMRI) will be used to assess intrinsic brain connectivity. Lower amplitude of low-frequency fluctuations (ALFF) and reduced functional connectivity (FC) within the default mode network (DMN) may reflect altered neural efficiency. Resting-state electroencephalography (rsEEG) will be employed to measure spontaneous neural oscillations. Enhanced theta/beta ratio and reduced alpha power may indicate compromised regulatory control and cortical arousal, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No